CLINICAL TRIAL: NCT04619602
Title: Pilot Study of an Inhaled Treatment for Bronchopulmonary Dysplasia
Brief Title: Inhaled Treatment for Bronchopulmonary Dysplasia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA hold
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Thomas Michael Raffay, MD, Sponsor-Investigator, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPD
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: bronchopulmonary dysplasia; respiratory failure
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GSNO therapy (Experimental): Intervention will be 30 minutes of inhaled GSNO agent in enrollment blocks of three subjects/dose (0.5 mL/kg of 0.25 mM, 0.5 mM, or 1 mM) to infants.
  Interventions: Drug: GSNO

INTERVENTIONS:
Drug: GSNO — Intervention will be 30 minutes of inhaled GSNO agent in enrollment blocks of three subjects/dose (0.5 mL/kg of 0.25 mM, 0.5 mM, or 1 mM) to infants.

SUMMARY:
The primary objective of this study is to provide expanded access of S-nitrosylation therapy for the treatment of bronchopulmonary dysplasia

DETAILED DESCRIPTION:
Open label study with 20 participants, open-label, with block dose escalation of 3 subjects/dose (0.5 mL/kg of 0.25 mM, 0.5 mM, or 1 mM). A minimum of seven days of surveillance will separate dosing blocks. An additional 11 subjects will be enrolled at the maximum 1 mM block (5x10-7 moles/kg). The primary outcomes are safety during 30 minutes of inhalation, and for 4 hours after inhalation, as measured by occurrence of adverse events related to the treatment + time period [during administration and tracked for next 7 days].

ELIGIBILITY:
Inclusion Criteria:

1. Inborn or outborn infants of either sex or any race or ethnicity
2. <32 weeks gestation at birth (best obstetrical dating)
3. Aged 29 to 365 days
4. Refractory hypoxic respiratory failure (average daily FiO2 >35% for 5 days)
5. Requires mechanical ventilation via endotracheal airway

Exclusion Criteria:

1. Life-threatening congenital or acquired anomalies (lethal chromosomal, thoracic/cardiac, brain)
2. Unstable condition defined as severe hypoxemia (FiO2 >85% for >24hrs), sepsis, or hypotension
3. Baseline methemoglobin > 3%, congenital methemoglobinemia, or a familial hemoglobinopathy
4. On steroid to facilitate endotracheal extubation
5. Individuals on inhaled nitric oxide, a phosphodiesterase 5 (PDE-5) inhibitor, taking allopurinol, β-adrenergic blockers, tricyclic antidepressants, meperidine (or related CNS agents), or nitrates
6. Thrombocytopenia defined as <50,000 platelets/µL on weekly NICU labs, clinical evidence of bleeding, on an anti-coagulant, or individuals with an inherited or acquired coagulation disorder
7. Anemia defined as a hemoglobin of < 9 mg/dL on weekly NICU labs
8. Concerns for pre-existing liver damage defined as an AST/ALT > 50 IU/L or direct bilirubin >1 mg/dL on weekly NICU labs
9. Concerns for acute kidney injury defined as a serum creatinine > 0.7 mg/dL on weekly NICU labs or 24-hr urine output <1.0 ml/kg/hr during preceding 4 days
10. Patients that are ventilated with a device not certified for blending of aerosolized solutions into the ventilator circuit
11. Physician of record opposed to enrolling the patient due to perceived safety concerns; or any condition that does not allow the protocol to be followed safely
12. Subjects that have experienced cardiac arrest with CPR for longer than 30 minutes

Ages: 29 Days to 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | 7 days
  Occurrence of >grade 3 adverse events related to the treatment

SECONDARY OUTCOMES:
S-nitrosoglutathione change | 30 minutes
  Percent change in S-nitrosoglutathione pre/post treatment
Change in oxygen saturation index | 4 hours
  Percent change in oxygen saturation index (O.S.I.) pre/post treatment. oxygen saturation index [O.S.I. = (FiO2) x (mean airway pressure) x 100 / (SpO2)]. High OSI scores indicate worse respiratory failure (high OSI = bad, low OSI = good).Scale range: zero - infinity
Change in GSNO catabolism pre/post treatment | 30 minutes
  Percent change in GSNO catabolism pre/post treatment
Intermittent hypoxemia as measured by oxygen saturation post treatment | 4 hours
  Incidence, duration, and nadirs of intermittent hypoxemia (SpO2 <80%) as measured by oxygen saturation parameters post treatment
Ventilator parameters post treatment | 4 hours
  Change in ventilator parameters post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Raffay, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No